CLINICAL TRIAL: NCT02530229
Title: Early Diagnostics of Septic Arthritis and Periprosthetic Joint Infections With Calorimetry and Polymerase Chain Reaction (PCR) of Synovial Aspirate Fluid
Brief Title: Arthrocentesis Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Berlin Institute of Health (Other)
Responsible Party: Principal Investigator, Andrej Trampuz, Head Septic Surgery Unit, Charite University, Berlin, Germany
Other Study IDs: EA1/306/14
Record Dates: First submitted 2015-08-19; First posted 2015-08-21 (Estimated); Last update posted 2015-08-21 (Estimated); Status verified 2015-08

CONDITIONS: Periprosthetic Joint Infection; Septic Arthritis
Keywords: periprosthetic joint infection; septic arthritis
MeSH Terms: conditions — Arthritis, Infectious

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples With DNA — joint aspirates of native joints and joints with suspected periprosthetic joint infection
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Periprosthetic joint infection: Patients with suspected periprosthetic joint infection of the hip, knee and shoulder
- Septic arthritis: Patients with suspected septic arthritis of a native joint of the hip, knee and shoulder

SUMMARY:
The purpose of this study is to analyze pre- and intra-operative joint aspirates of native joints and joints with suspicion of periprosthetic joint infection (PJI) of the hip, knee and shoulder acquired in clinical routine. Joint aspirates are then analyzed with new diagnostic methods (microcalorimetry, PCR, alpha-defensin, etc.). Diagnostic speed and accuracy of these methods is compared to standard diagnostic methods in clinical routine, such as blood cultures of joint aspirates, cell count/differential, intra-operative tissue culture and histology and sonication.

DETAILED DESCRIPTION:
In this study, joint aspirate of patients that undergo joint aspiration in the context of routine pre- and intra-operative clinical diagnosis of a hip, knee or shoulder joint is collected. Routine joint punctures at our clinic are regularly performed in the emergency room, in the outpatient clinic and intra-operatively during diagnostic and revision surgery. A minimum of 5 ml aspiration fluid was required for inclusion in this study. Empty or diluted aspirations were excluded.

Joint aspirations are performed by orthopaedic surgeons with an 18-gauge needle according to standardized aseptic technique. Intraoperative punctures are performed prior to arthrotomy. A minimum of 1ml of joint aspirate is immediately transferred to a native study vial for our study, a native vial for gram stain and culture and a native vial for polarization microscopy, respectively. A minimum of 1 ml joint aspirate is transferred to an ethylenediaminetetraacetic acid (EDTA) vial for the determination of leucocyte count. Finally, a minimum of 1 ml is inoculated into a paediatric blood culture bottle.

Standard microbiological methods are performed in an external laboratory that routinely collaborates with our clinic. Leucocyte count is performed automatically with the mentioned EDTA vial. Polarization microscopy is performed at our pathohistological department in order to detect crystals and signs of infection in joint aspirate.

If written informational consent has been signed by the patient, the study vial is immediately transported to our internal laboratory for analysis with new diagnostic methods (microcalorimetry, PCR, etc.). When an immediate transportation was not feasible, the vial is stored in a cooling fridge at +3° C until transportation was possible.

Each case is individually reviewed and classified by an experienced infectiologist taking the case's clinical history and laboratory results into account.

ELIGIBILITY:
Inclusion Criteria:

* adult of 18 or more years
* written consent to participate in study
* suspicion of septic arthritis or periprosthetic joint infection
* joint aspirate minimum of 5 ml

Exclusion Criteria:

* is not able to understand the aim or purpose of this study
* empty joint aspirate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient with suspicion of septic arthritis or periprosthetic joint infection of the hip, knee and shoulder being diagnosed or treated in our facility in a clinical routine scenario willing to participate in this study (written informational consent)
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2014-11; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
growth of microbial agent in culture of joint aspirate | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Andrej Trampuz, MD, Principal Investigator — Charité University Berlin
Locations (1):
- Charité University Berlin, Berlin, State of Berlin, Germany

REFERENCES:
- [Background] Yusuf E, Hugle T, Daikeler T, Voide C, Borens O, Trampuz A. The potential use of microcalorimetry in rapid differentiation between septic arthritis and other causes of arthritis. Eur J Clin Microbiol Infect Dis. 2015 Mar;34(3):461-5. doi: 10.1007/s10096-014-2248-y. Epub 2014 Sep 25. PMID 25252631
- [Background] Corvec S, Portillo ME, Pasticci BM, Borens O, Trampuz A. Epidemiology and new developments in the diagnosis of prosthetic joint infection. Int J Artif Organs. 2012 Oct;35(10):923-34. doi: 10.5301/ijao.5000168. PMID 23138706
- [Background] Trampuz A, Hanssen AD, Osmon DR, Mandrekar J, Steckelberg JM, Patel R. Synovial fluid leukocyte count and differential for the diagnosis of prosthetic knee infection. Am J Med. 2004 Oct 15;117(8):556-62. doi: 10.1016/j.amjmed.2004.06.022. PMID 15465503
- [Background] Zimmerli W, Trampuz A, Ochsner PE. Prosthetic-joint infections. N Engl J Med. 2004 Oct 14;351(16):1645-54. doi: 10.1056/NEJMra040181. No abstract available. PMID 15483283
- [Derived] Karbysheva S, Cabric S, Koliszak A, Bervar M, Kirschbaum S, Hardt S, Perka C, Trampuz A. Clinical evaluation of dithiothreitol in comparison with sonication for biofilm dislodgement in the microbiological diagnosis of periprosthetic joint infection. Diagn Microbiol Infect Dis. 2022 Jun;103(2):115679. doi: 10.1016/j.diagmicrobio.2022.115679. Epub 2022 Mar 12. PMID 35395437
- [Derived] Morgenstern C, Renz N, Cabric S, Maiolo E, Perka C, Trampuz A. Thermogenic diagnosis of periprosthetic joint infection by microcalorimetry of synovial fluid. BMC Musculoskelet Disord. 2020 Jun 3;21(1):345. doi: 10.1186/s12891-020-03366-3. PMID 32493292
- [Derived] Sigmund IK, Renz N, Feihl S, Morgenstern C, Cabric S, Trampuz A. Value of multiplex PCR for detection of antimicrobial resistance in samples retrieved from patients with orthopaedic infections. BMC Microbiol. 2020 Apr 14;20(1):88. doi: 10.1186/s12866-020-01741-7. PMID 32290833
- [Derived] Morgenstern C, Renz N, Cabric S, Perka C, Trampuz A. Multiplex Polymerase Chain Reaction and Microcalorimetry in Synovial Fluid: Can Pathogen-based Detection Assays Improve the Diagnosis of Septic Arthritis? J Rheumatol. 2018 Nov;45(11):1588-1593. doi: 10.3899/jrheum.180311. Epub 2018 Sep 15. PMID 30219763